CLINICAL TRIAL: NCT02255877
Title: A Prospective, Non Blinded, Randomized Controlled Post Market Study Designed to Compare the Use of the Zip Surgical Skin Closure Device vs. Conventional Steel Staples for Skin Closure in Subjects Who Undergo a bi Lateral Knee Arthroplasty
Brief Title: ZIPS Study - Zip Incision Approximation vs. STAPLE
Acronym: ZIPS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in research plan
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Bi lateral knee surgery; uni compartmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zip Surgical Skin Closure (Active Comparator): Subjects randomized to receive one knee (left or right) closed with ZipSurgical Skin Closure and the other knee closed with standard staples
  Interventions: Device: Zip Surgical Skin Closure; Device: Steel Staples
- Steel Staples (Active Comparator): Subjects randomized to receive one knee (left or right) closed with Staples and the other knee closed with ZipSurgical Skin Closure
  Interventions: Device: Zip Surgical Skin Closure; Device: Steel Staples

INTERVENTIONS:
Device: Zip Surgical Skin Closure — Non invasive skin closure device for closure of the skin layer for surgical incisions or laceration repair.
  Other Names: Zip 16; Zip 8i
Device: Steel Staples — Skin Closure device for the closure of the skin layer for surgical incisions.

SUMMARY:
Study designed to evaluate the Zip Surgical Skin Closure device versus conventional steel staple placement when utilized for surgical wound closure after bi lateral unicompartmental or bi later total knee replacement.

DETAILED DESCRIPTION:
This is a randomized, within patient control study aiming to enroll up to 25 subjects requiring bi lateral knee arthroplasty (unicompartmental or toal) at a single study center. Subjects will be followed for up for 6 weeks post surgery to evaluate wound healing and overall satisfaction of closure methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring epidermal closure after bi lateral total or partial (unicompartmental) knee arthroplasty;
* Patients willing to be evaluated at discharge and 6-weeks post op.

Exclusion Criteria:

* Known bleeding disorder not caused by medication
* Known personal or family history of keloid formation or scar hypertrophy
* Known allergy or hypersensitivity to non-latex skin adhesives
* Atrophic skin deemed clinically prone to blistering
* Any skin disorder affecting wound healing
* Any other condition that in the opinion of the investigator would make a particular patient unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness Outcome - Wound Healing | 6 weeks post surgery
  Wound healing as judged by the Cosmetic Visual Analogue Scale - Photos taken at 6 weeks post surgery will be judged by panel of Plastic Surgeons blinded to the treatment assignments.

SECONDARY OUTCOMES:
Surgeon Satisfaction with the Closure Method | At Discharge, 1-3 days post surgery
  Closure Method satisfaction (Zip and Staple) will be collected with a 5 point satisfaction scale (from very satisfied to very dissatisfied)
Patient Pain | Throughout 6 week study period (Discharge, 2 week follow up and 6 week follow up (exit) visits.)
  General post operative and incisional pain levels will be collected using a 10 point VAS scale
Patient Satisfaction of Scars | At 6 week Follow up (exit) visit
  Scar satisfaction (Zip and Staple) will be collected with a 5 point satisfaction scale (from very satisfied to very dissatisfied) and with a 10 point VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storne, Study Director — VP Marketing
Locations (1):
- Orthopaedic Research Foundation, Indianapolis, Indiana, United States